CLINICAL TRIAL: NCT02456454
Title: Placebo Controlled Trial of Valproate Versus Risperidone in Young Children With Bipolar Disorder
Brief Title: Controlled Trial of Valproate Versus Risperidone in Young Children With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Robert Kowatch, MD, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHMC#03-12-26
Record Dates: First submitted 2015-04-24; First posted 2015-05-28 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Risperidone (Experimental): Risperidone, PO 0.25-2 mg/day
  Interventions: Drug: Risperidone
- Valproic (Experimental): Valproic Acid PO to achieve plasma levels of 85-100
  Interventions: Drug: Valproic Acid
- Placebo (Placebo Comparator): Liquid placebo PO matched for color and taste.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — Liquid risperidone
  Other Names: Risperdal
  Arms: Risperidone
Drug: Valproic Acid — Liquid valproic acid
  Other Names: Valproate
  Arms: Valproic
Drug: Placebo
  Arms: Placebo

SUMMARY:
Controlled trial of the efficacy and safety of valproate, versus risperidone in children, ages 3-7 yr. with Bipolar I or II Disorder, mixed, manic or hypomanic episode.

DETAILED DESCRIPTION:
The objective of this study was to study the efficacy and safety of valproate, versus risperidone in children, ages 3-7 yr. with Bipolar I or II Disorder, mixed, manic or hypomanic episode.

ELIGIBILITY:
Inclusion Criteria

* Subjects were male or female outpatient subjects,
* 3.0 - 7 years 11 months of age
* Bipolar I or II Disorder, mixed, manic or hypomanic episode, psychotic or non-psychotic, according to DSM IV criteria (American Psychiatric Association 1994)
* with a score > 20 on the Young Mania Rating Scale (YMRS.

Exclusion Criteria

* clinically significant or unstable hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrinologic, immunologic, hematologic or other systemic medical conditions;
* neurologic disorders including epilepsy, stroke, or severe head trauma those clinically significant laboratory abnormalities, on any of the following tests:

  * CBC with differential,
  * electrolytes,
  * BUN,
  * creatinine,
  * hepatic transaminases,
  * urinalysis,
  * thyroid indices (T3, Total T4, Free T4, TSH) and
  * EKG
* mania due to a general medical condition or substance-induced mania
* mental retardation (IQ <70),
* evidence of Fetal Alcohol Syndrome or an Alcohol-Related Neurodevelopmental Disorder,
* Schizophrenia or other psychotic disorders (including schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale | 6 weeks
  Young Mania Rating Scale

SECONDARY OUTCOMES:
Clinical Global Improvement Scale | 6 weeks
  Clinical Global Improvement Scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Kowatch, MD, PhD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kowatch RA, Scheffer RE, Monroe E, Delgado S, Altaye M, Lagory D. Placebo-controlled trial of valproic Acid versus risperidone in children 3-7 years of age with bipolar I disorder. J Child Adolesc Psychopharmacol. 2015 May;25(4):306-13. doi: 10.1089/cap.2014.0166. PMID 25978742